CLINICAL TRIAL: NCT00002220
Title: Multi-Center, Open-Label Study of the Effect of Indinavir, Efavirenz, and Adefovir Dipivoxil Combination Therapy in Patients Who Have Failed Nelfinavir
Brief Title: Indinavir Plus Efavirenz Plus Adefovir Dipivoxil in HIV-Infected Patients Who Have Not Had Success With Nelfinavir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246N; 075-00; NCT00002242 (obsolete NCT alias)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Drug Resistance; Drug Therapy, Combination; Antiviral Agents; HIV Protease Inhibitors; Indinavir; RNA, Viral; Adenine; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; efavirenz; Carnitine; adefovir dipivoxil

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Efavirenz
Drug: Levocarnitine
Drug: Adefovir dipivoxil

SUMMARY:
The purpose of this study is to compare the effectiveness of giving indinavir plus efavirenz plus adefovir dipivoxil to patients who have failed treatment with nelfinavir and patients who have never taken a protease inhibitor (PI). Effectiveness is measured by the number of patients who have a viral load (level of HIV in the blood) below 400 copies/ml after 48 weeks of treatment.

DETAILED DESCRIPTION:
In this open-label, nonrandomized study, 120 HIV-infected patients are stratified into two groups: failed nelfinavir vs protease inhibitor-naive. All patients receive indinavir plus efavirenz plus adefovir dipivoxil plus and L-carnitine, orally. Plasma vRNA is measured every 4 weeks until Week 16, then every 8 weeks for the remainder of the 48-week study.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serologically documented HIV infection.
* Baseline CD4 count greater than or equal to 50 cells and vRNA greater than or equal to 10,000 copies/ml.
* Parental consent for patients under 18.

Nelfinavir-Failure Group:

* Must have protease inhibitor experience solely with nelfinavir and be considered drug-adherent.
* Must be candidate for changing therapy because of virologic failure and be receiving nelfinavir at entry (at least 16 weeks of nelfinavir plus NRTI therapy with at least a 10-fold decline in vRNA due to nelfinavir therapy and a subsequent increase toward the patient's baseline vRNA of at least 10-fold).

Control Group:

* Must have received any combination of currently licensed nucleoside reverse transcriptase inhibitors for at least 16 weeks.
* Must be naive to efavirenz, adefovir dipivoxil, and other NRTI's.

Exclusion Criteria

Prior Medication:

Excluded:

Control group:

* Prior efavirenz, adefovir dipivoxil, or other non-nucleoside reverse transcriptase inhibitors.

Required:

Nelfinavir-failure patients:

* At least 16 weeks of nelfinavir.

Control group:

* At least 16 weeks of any combination of currently licensed nucleoside reverse transcriptase inhibitors.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - LAC / USC Med Ctr / Infectious Diseases, Los Angeles, California
  - Yale Univ / AIDS Clinical Trials Unit, New Haven, Connecticut
  - Med Ctr of Delaware, Wilmington, Delaware
  - Hawaii AIDS Clinical Trial Unit, Honolulu, Hawaii
  - Rush Presbyterian Saint Lukes Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Columbia Presbyterian Hosp, New York, New York
  - AIDS TMT Unit / Univ Hosp, Stony Brook, New York
  - Vanderbilt Clinic, Nashville, Tennessee
  - Oaklawn Physicians Group, Dallas, Texas